CLINICAL TRIAL: NCT04684771
Title: Evaluation of Efficacy and Tolerance of a Food Supplement (MYOSTIM®) in Postoperative Revalidation of Patients After Reconstructive Surgery of Anterior Cruciate Ligament
Brief Title: Tolerance, Efficacy, revAlidation, Myostim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alternativa International S.A (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TEAM
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: food supplement; revalidation after surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Double blind, exploratory study, monocentric, with a group of control patient with placebo.
  Two parallel-groups receiving during 12 weeks either the MYOSTIM® or a PLACEBO in a double blinded manner.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two parallel-groups either the MYOSTIM® or a PLACEBO in a double blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MYOSTIM® (Active Comparator): MYOSTIM® 2 bars/day during 12 weeks MYOSTIM® as a food bar. Active ingredient: Pomegranate extract, L-leucine, Creatine, D3 Vitamin, Proteins IP Status: Food supplement n° NCT 2485/8 (Red fruits flavor bar) and NCT 2485/7 (Black chocolate flavor bar) delivered by the Federal Public Service, Health, Food chain safety and environment.
  Interventions: Dietary Supplement: MYOSTIM®
- PLACEBO (Placebo Comparator): PLACEBO 2 bars/day during 12 weeks
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: MYOSTIM® — Food supplement n° NCT 2485/8 (Red fruits flavor bar) and NCT 2485/7 (Black chocolate flavor bar) delivered by the Federal Public Service, Health, Food chain safety and environment.
  Arms: MYOSTIM®
Dietary Supplement: PLACEBO — Bars with no active ingredient and the same flavor (chocolate and red fruits).
  Arms: PLACEBO

SUMMARY:
Evaluation of efficacy and tolerance of a food supplement (MYOSTIM®) versus a placebo in postoperative revalidation of patients after reconstructive surgery of anterior cruciate ligament.

The food supplement (MYOSTIM®) has been developped and is supplied as food bars and composed of pomegranate, leucine, creatine, proteins and D vitamin. The aim of this exploratory study is to assess the efficacy and tolerance of MYOSTIM® on muscle performance after ACL reconstructive surgery and in postoperative revalidation phase.

ELIGIBILITY:
Inclusion Criteria:

* Male between the age of 18 and 40
* BMI (Body Mass Index) ≤ 27
* Candidates for ACL reconstruction surgery of DIDT (Droit Interne et du Demi Tendineux) type
* Able to follow the instruction of the study, to go to the postoperative visits to the investigator, to go to the isokinetic and to the MRI visits
* Having signed an informed consent

Exclusion Criteria:

Related to the pathology:

* Patient who have undergone previous ACL reconstruction surgery on the same knee
* Patient who have participated to a therapeutic clinical study 3 months before inclusion
* Patient who plan to follow a workout or a revalidation program after surgery different from classical physiotherapy prescribed by the orthopedic surgeon
* Contralateral limb suffered from trauma, surgery, fracture, tear, tendinopathy, sepsis or immobilization for more than 3 weeks during the last 5 years

Related to treatment:

* Patient who have eaten doping substances or food supplement building mass and muscle strength during 3 months before inclusion excepted for creatine and beta-alanine for which the washout period is of 6 month before inclusion
* Patient who were treated with antibiotics in the month preceding the inclusion
* Patient treated with pharmacologic agents like statins, immunosuppressors or anti-malaria
* Patient taking androgens (steroids…)
* Patient under treatments which may interfere with the neuromuscular system
* Patient who were treated with analgesic or non-steroidal anti-inflammatory drugs (NSAIDS) 24 hours before inclusion visit

Related to associated diseases:

* Patient with associated uncontrolled severe disease: severe liver or kidney disease, severe and uncontrolled cardiovascular disease, HIV, B or C hepatitis, tumor
* Patient with thromboembolism disorders
* Patient with inflammatory bowel disease
* Anorexic patient
* Diabetic patient
* Patient with traumatic, neurologic or rheumatic history of the lower limbs

Related to patient:

* Allergy or contraindication to soy, milk, gluten, nuts or wheat
* Forecasting a high protein diet during the study
* Under guardianship or judicial protection

Related to MRI counter-indication:

* Patient with a pacemaker, an implantable defibrillator, neurosurgical clips, a neurostimulator, cochlear implant, a stent from less than 3 weeks, an insulin pump
* Patient with a ferromagnetic splinter in the body, or having wire sutures
* Serious mobility problem (Parkinson, tremors)
* Claustrophobia

Related to impedancemeter test:

• Patient with a metal plate at the right ankle

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of MYOSTIM® on the muscular strength recovery | Change from Baseline at 14 weeks post ACL surgery
  Evaluation by isokinetic test performed (extension/flexion of the quadriceps)
Assess the efficacy of MYOSTIM® on the muscular strength recovery | Change from Baseline at 14 weeks post ACL surgery
  Evaluation by isokinetic test performed (extension/flexion of the hamstrings)
Assess the efficacy of MYOSTIM® on the muscular mass recovery | Change from Baseline at 14 weeks post ACL surgery
  Evaluation by Magnetic Resonance Imaging (MRI)
Assess the efficacy of MYOSTIM® on the muscular mass recovery | Change from Baseline at 14 weeks post ACL surgery
  Evaluation by impedancemetry
Assess the efficacy of MYOSTIM® on physical performance recovery | Change from Baseline at 14 weeks post ACL surgery
  Evaluation with one self-administrated knee evaluation questionnaire from the International Knee Documentation Committee
Assess the effect of MYOSTIM® on blood biomarker | Change from Baseline at 2 and14 weeks post ACL surgery
  Evaluation of blood concentration of biomarker (Myostatin (muscular atrophy), Myeloperoxidase (chronic joint inflammation), Coll2-1 and Coll2-1NO2 (Cartilage inflammation and degradation), IL6 (muscular atrophy and inflammation), MMP3 and NT-CAF (cartilage and neuro-muscular junction), TNFa (inflammation))
Assess the efficacy of MYOSTIM® on the pain of the patient | Change from Baseline at 2 and14 weeks post ACL surgery
  Evaluation of pain of the patient by one visual analogue scale (VAS)
Assess the efficacy of MYOSTIM® on the global judgment of the patient | Change from Baseline at 2 and14 weeks post ACL surgery
  Evaluation of global judgment of the patient by one visual analogue scale (VAS)
Assessment of the tolerance of the patient with the MYOSTIM® | At 14 weeks post ACL surgery
  Evaluation according the number of Adverse Events (AE), remaining bars and satisfaction scale for the product
Assessment of the compliance of the patient with the MYOSTIM® | At 14 weeks post ACL surgery
  Evaluation according the number of remaining bars
Assessment of the satisfaction of the patient with the MYOSTIM® | At 14 weeks post ACL surgery
  Evaluation according the satisfaction scale for the product

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Hospital Bois de l'Abbaye et de Hesbaye, Seraing, Liège
  - CHU de Liège, Liège